CLINICAL TRIAL: NCT00457587
Title: Präklinische Studie Zur Etablierung Einer Immuntherapie für Das Nebennierenrindenkarzinom - Preclinical Study Towards an Immunotherapy in Adrenocortical Carcinoma
Brief Title: Preclinical Study Towards an Immunotherapy in Adrenocortical Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wuerzburg (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Martin Fassnacht, Professor for Internal Medicine and Endocrinology, University of Wuerzburg
Other Study IDs: Wue-Immuno-ACC-83/05
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Adrenocortical Carcinoma; Cushing's Syndrome
MeSH Terms: conditions — Adrenocortical Carcinoma; Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — whole blood for monocytes isolation serum urine tumor samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Adrenocortical carcinoma (ACC) is a rare and heterogeneous malignancy with poor prognosis. Surgical resection of the tumor is the treatment of choice. However, even after complete resection more than 80 % of patients will experience recurrence of disease. Therefore, new treatment options are urgently needed. This pre-clinical study try to lay the foundations for a successful immunotherapy in patients with ACC.

ELIGIBILITY:
Inclusion Criteria:

* patients with histological proven adrenocortical carcinoma
* healthy persons as control group
* Life expectancy > 6 months

Exclusion Criteria:

* autoimmune diseases
* severe clinical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adrenocortical carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To find reasonable antigens for a vaccination therapy in ACC | day of blood sampling
To investigate the role of tumor-induced suppression in ACC | NA, in vitro study

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fassnacht, MD, Principal Investigator — University of Wuerzburg
Locations (1):
- Dept. of Medicine I, University of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Result] Landwehr LS, Altieri B, Schreiner J, Sbiera I, Weigand I, Kroiss M, Fassnacht M, Sbiera S. Interplay between glucocorticoids and tumor-infiltrating lymphocytes on the prognosis of adrenocortical carcinoma. J Immunother Cancer. 2020 May;8(1):e000469. doi: 10.1136/jitc-2019-000469. PMID 32474412
- See also: Homepage Dept. of Endocrinology, U Wuerzburg — https://www.ukw.de/medizinische-klinik-i/endokrinologie/startseite/